CLINICAL TRIAL: NCT03812367
Title: Prospective Study to Assess Changes in the Number and Activity of Pre-Osteoclasts and Osteoclasts Over Time in Postmenopausal Women Treated With Denosumab or Zoledronic Acid
Brief Title: Activity of Pre-Osteoclasts and Osteoclasts Over Time in Postmenopausal Women Treated With Denosumab or Zoledronic Acid
Status: Withdrawn | Type: Observational
Why Stopped: The Investigator decided not to pursue this study.
Sponsor: University of California, Davis (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 1030286
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: The denosumab naïve group
- Group 2: The zoledronic acid naïve group
- Group 3: The chronic denosumab (> 1 year with at least 3 biannual injections)
- Group 4: The chronic zoledronic acid (≥2 years with at least 2 annual injections)

SUMMARY:
This study evaluates how patients treated with denosumab or zoledronic acid for osteoporosis may change the number of peripheral osteoclast precursors and osteoclast activity, and how that may be associated with changes in bone mass.

DETAILED DESCRIPTION:
Postmenopausal osteoporosis is the leading cause of low trauma fractures. At the time of menopause there is an uncoupling of bone turnover, with osteoclast mediated bone resorption increased more than bone formation, resulting in both loss of bone mass and architecture such that bone fractures with very little force.

Bisphosphonates are commonly used to treat postmenopausal osteoporosis, although the mechanisms of their action on bone are not completely understood. Gossiel and colleagues recently examined the effects of ibandronate, alendronate and risedronate on osteoclast precursor cells in a study of women (n=62) with postmenopausal osteoporosis. Fasting serum was collected at baseline and after 1 and 48 weeks of bisphosphonate treatment. Fluorescent-activated cell sorting (FACS)-Calibur was used to extract peripheral blood mononuclear cells (PBMC), and cells were stained for receptors of macrophage colony stimulating factor (M-CSFR) and tumor necrosis factor 2 (TNFR2), as well as adhesion molecules (CD11b and CD14). These cell surface antigens are important for osteoclast differentiation and activity. Osteoclast precursor cells were identified using flow cytometry to find cells that were dual positive (CD14+/M-CSFR+, CD14+/CD11b+, CD14+/TNFR2+). Results showed a significant (p<0.01) reduction in in expression of M-CSFR (53% decrease) and CD11b (49% decrease) after 48 weeks of treatment, suggesting that the action of bisphosphonates on mature osteoclasts may be mediated by reduction of osteoclast precursor cells.

Treatment with denosumab (a monoclonal antibody that blocks the ability of receptor activator of NFκB ligand [RANKL] to bind to its receptor RANK on the osteoclast surface and inhibits the maturation and activity of osteoclasts) has been found to increase bone mineral density (BMD) at the lumbar spine and hip in both postmenopausal women and elderly men with osteopenia. However, after denosumab is discontinued there can be a rapid loss of BMD and an increased incidence of vertebral fractures. Current data suggests that the incidence of vertebral fracrure increases to levels similar to placebo after denosumab discontinuation, and only the incidence of multiple vertebral fracture is higher after denosumab discontinuation compared with placebo discontinuation, though further research is needed. The increase in the observed bone loss may be from increased osteoclast maturation and activity, or an change in the number circulating monocytes (the precursors of osteoclasts) during the denosumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women at least 50 years of age who are postmenopausal. Postmenopausal is defined as being amenorrheic for at a period of at least 12 months.
2. Diagnosis of osteoporosis by T score of < -2.5 at either lumbar spine or the hip/femoral neck, or osteopenia that qualifies for treatment by FRAX calculation (10-year risk of hip fracture > 3% and/or major osteoporotic fracture of > 20%).

3a. Subjects who have had chronic treatment of denosumab (as defined as > 1 year [at least 3 6-monthly injections]) or zoledronic acid (defined as ≥ 2 years [at least 2 annual injections]) . Note: At the time of treatment initiation, subjects must have met criteria for on-label use (e.g. criterion 2 above).

OR 3b. Subjects who are naïve to treatment with denosumab and/or zoledronic acid.

Exclusion Criteria:

1. Renal insufficiency, with glomerular filtration rate (GFR) < 35 ml/min.
2. Hypocalcemia within 6 months of study initiation.
3. Known hypersensitivity to denosumab or zoledronic acid.
4. Medications that could alter bone turnover including prednisone, anti-rheumatic medications, anti-metabolites (Cytoxan). Subjects who have been on stable doses of thyroid replacement or diabetes medications for more than 3 months are eligible.
5. Evidence of untreated oral cavities or oral infections. Preventative dental exams should be performed before starting denosumab or zoledronic acid. Subjects must avoid invasive dental procedures during treatment with denosumab or zoledronic acid.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged > 50 with diagnosis of osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in osteoclast circulation | 1 month, 6 months, 12 months
  Percent change (%Δ) from baseline in number of circulating osteoclast precursor cells by FACS analysis
Percent change in osteoclast maturation and activity | 1 month, 6 months, 12 months
  Percent change (%Δ) in osteoclast maturation and activity, as assessed by resorption on dentin slides and expression of genes critical for osteoclast differentiation
Percent change in number of TRAP cells | 1 month, 6 months, 12 months
  Percent change (%Δ) from baseline in the number of tartrate-resistant acid phosphatase (TRAP)+cells with 3 or mor nuclei by in vitro maturation
Percent change in bone mass density | 1 month, 6 months, 12 months
  Percent change (%Δ) from baseline in BMD at the total hip and lumbar spine
Percent change in bone turnover markers | 1 month, 6 months, 12 months
  Percent change (% Δ) from baseline in bone turnover markers C-telopeptide of type 1 collagen (CTX) and procollagen type 1 propeptide (P1NP)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lane, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Health, Center for Musculoskeletal Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided